CLINICAL TRIAL: NCT01090440
Title: An Open Label, Randomised, Three-way Cross-over Study to Evaluate the Pharmacokinetics, Effect of Food, Safety and Tolerability of a New Tablet Formulation of GSK1144814 in Healthy Male and Female Subjects
Brief Title: Pharmacokinetics, Effect of Food, Safety and Tolerability of a New Tablet Formulation of GSK1144814 in Healthy Subjects
Acronym: MNK112891
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 112891
Record Dates: First submitted 2010-03-04; First posted 2010-03-22 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia; GSK1144814; effect of food; healthy subjects; depressive disorder; pharmacokinetics
MeSH Terms: conditions — Schizophrenia; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Three-way cross- over (Experimental): Three regimens will be administered in this study: A: GSK1144814 Tablet (100mg) Fasted State; B: GSK1144814 Tablet (200mg) Fasted State and C: GSK 1144814 Tablet (100mg) Fed State (FDA high fat breakfast).
  Interventions: Drug: GSK1144814

INTERVENTIONS:
Drug: GSK1144814 — This study is an open label, randomised, three-way cross-over study to evaluate the pharmacokinetics, effect of food, safety and tolerability of a new tablet formulation of GSK1144814 in healthy male and female (non-child bearing potential) subjects. Sixteen subjects will be enrolled to provide a minimum number of 12 evaluable subjects. The doses to be administered will be 100 mg and 200mg in the fasted state, and 100mg following a high fat breakfast.

SUMMARY:
GSK1144814 is a potent, insurmountable antagonist at human neurokinin-1 (NK1) and neurokinin-3 (NK3) receptors with the potential to treat multiple symptom domains of schizophrenia and be an efficacious antidepressant.

This study will be an open label, randomised, three-way cross-over study to evaluate the safety, tolerability and pharmacokinetics of a new tablet formulation of GSK1144814 and to evaluate the effect of food on single oral doses of GSK1144814 in healthy male and female subjects.

DETAILED DESCRIPTION:
GSK1144814 is a potent, insurmountable antagonist at human neurokinin-1 (NK1) and neurokinin-3 (NK3) receptors with the potential to treat multiple symptom domains of schizophrenia and be an efficacious antidepressant.

This study will be an open label, randomised, three-way cross-over study to evaluate the safety, tolerability and pharmacokinetics of a new tablet formulation of GSK1144814 and to evaluate the effect of food on single oral doses of GSK1144814 in healthy male and female (non-child bearing potential) subjects.

The study will consist of a Screening visit (up to 30 days before the first dosing session), three dosing sessions each separated by a maximum of at least 6 days washout, and a Follow up visit (7 to 14 days after the last dose of study medication). Each subject's participation in the study will be approximately 12 weeks Sixteen subjects will be enrolled to provide a minimum number of 12 evaluable subjects. The doses to be administered will be 100 mg and 200mg in the fasted state, and 100mg following a high fat breakfast.

Subjects will be admitted to the unit on Day 1 of each dosing session and will remain in the unit until 48 hours after dosing. Pharmacokinetic samples will be taken for up to 72 hours post dose. The duration of both in patient stay and PK sampling may be subject to change depending on emerging safety and PK results. Dosing will be in the morning approximately the same time for all sessions.

The objectives of the study are to evaluate the pharmacokinetics, safety and tolerability of GSK1144814. Pharmacokinetic objectives are to evaluate the pharmacokinetic parameters of single oral doses of GSK1144814 administered as a tablet formulation in healthy male and female subjects and to evaluate the effect of a high-fat meal on the pharmacokinetics of GSK1144814 tablet following single dose administration of GSK1144814 to healthy male and female subjects.

The safety and tolerability objectives are to evaluate the safety and tolerability of single oral doses of GSK1144814 tablet formulation in fed and fasted states.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinically significant abnormality or laboratory parameters significantly outside the reference range for the population being studied may be included only if the Investigator and the and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age.
* A female subject is eligible to participate if she is of:

Non childbearing potential defined as pre menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] greater than 40 mIU/mL and oestradiol less than 40 pg/mL [less than 140 pmol/L] is confirmatory).

Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to discontinue HRT to allow confirmation of post menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

* Male subjects must agree to use one of the contraception methods alloed by the protocol. This criterion must be followed from the first dosing day until 3 months after the last dose.
* Body weight greater than or equal to 50 kg and BMI within the range 19 to 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Demonstrates no evidence of mental impairment or co-morbid psychiatric disorders

Exclusion Criteria:

* History or presence of clinically significant cardiac arrhythmias, or other clinically significant cardiac disease.
* QTcB or QTcF greater than 450 msec.
* Subjects, who in the investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 6 months.
* The subject has a positive pre study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre study hepatitis B surface antigen (HBsAg) or positive hepatitis C virus (HCV) antibody test result within 3 months of Screening.
* A positive test result for antibodies to human immunodeficiency virus (HIV) 1/2.
* Significant renal abnormality (from medical history or as indicated by laboratory investigations). Additionally subjects with idiopathic haematuria or proteinuria or conditions such as benign orthostatic proteinuria and benign familial haematuria should be excluded from the study.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine containing products within 6 months prior to Screening.
* Subjects, who in the investigator's judgement, pose a significant homicidal risk or have ever been homicidal.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as the following Australian guidelines:

An average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to 270ml of full strength beer, 470ml of light beer, 30ml of spirits and 100ml of wine.

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Consumption of Seville oranges (including marmalade) and/or grapefruit and/or Chinese grapefruit (pomelo) and/or grapefruit hybrids and/or exotic citrus fruits and/or their fruit juices from 7 days prior to the first dosing day.
* Consumption of red wine from 7 days prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2009-10-09 (Actual); Study Completion 2009-10-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: tlag, Cmax, tmax, AUC(0-24), AUC(0 t), t½ and AUC(0 to infinity). | 2 months

SECONDARY OUTCOMES:
Safety and tolerability: AE monitoring, vital signs (blood pressure, heart rate, body temperature, electrocardiograms (ECGs) (12 lead and Holter), clinical laboratory assessments (standard laboratory parameters). | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- See also: Results for study 112891 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112891?search=study&study_ids=112891#rs